CLINICAL TRIAL: NCT01101529
Title: A Randomized Controlled Study to Compare (EMEND®)to Standard Treatment as Prevention for Delayed Chemotherapy-induced Nausea and Vomiting (CINV) After Myeloablative Therapy for Patients Undergoing Autologous Stem Cell Transplantation.
Brief Title: Treatment of Chemotherapy-induced Nausea and Vomiting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Gunnar Birgegard, Prof, Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EudraCT nr: 2009-010545-31; 2009-010545-31 (EudraCT Number)
Record Dates: First submitted 2010-04-09; First posted 2010-04-12 (Estimated); Last update posted 2012-12-13 (Estimated); Status verified 2012-12

CONDITIONS: Nausea; Vomiting
Keywords: Chemotherapy-induced nausea and vomiting CINV
MeSH Terms: conditions — Nausea; Vomiting | interventions — Aprepitant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard antiemetic therapy plus placebo (Placebo Comparator): Standard anti-emetic prophylaxis consisting of 1/dexamethasone 6 mg daily during the chemotherapy days and 2/tropisetron (Navoban)5 mg daily during chemotherapy and 2 days after
  Interventions: Drug: Placebo
- aprepitant (Emend) (Experimental): Aprepitant given orally 125 mg the first day, then 80 mg daily during the chemotherapy course and 7 days after as an addition to standard antiemetic therapy as in the placebo arm.
  Interventions: Drug: Aprepitant (Emend)

INTERVENTIONS:
Drug: Aprepitant (Emend) — Aprepitant will be added to the standard anti-emetic therapy. Emend is given orally, 125 mg the first day, then 80 mg daily during the chemotherapy course and 7 days after
  Other Names: Emend
  Arms: aprepitant (Emend)
Drug: Placebo — Placebo will be administered instead of Emend
  Arms: Standard antiemetic therapy plus placebo

SUMMARY:
Delayed nausea is a common problem after high dose chemotherapy for bone marrow transplantation. This study wants to compare standard prophylactic anti-emetic therapy with the same treatment plus the drug aprepitant (Emend). The hypothesis is that addition of Emend will reduce nausea and vomiting.

DETAILED DESCRIPTION:
A single centre randomized placebo-controlled phase II-study with a random assignment to experimental (EXP) or control (CTR) group. All patients with lymphoproliferative diseases ≥18 years of age, scheduled for myeloablative therapy before autologous stem cell transplantation at the Akademiska University Hospital in Uppsala, Sweden, will be included consecutively during one and a half year. A total of 90 patients (45 per treatment arm) will be accrued for this study. They will be invited by mail to participate in the study a couple of weeks before hospital entry. A random assignment to EXP or CTR will be performed by research nurses not participating in any other way in the study. Patients will be stratified for diagnosis which also means myeloablative therapy (lymphoma (BEAC) or myeloma (high-dose melphalan)), and the groups are expected to be similar in size. One box for each diagnosis (lymphoma and myeloma) will contain equal numbers of randomisation cards for the experimental and control groups, randomly mixed within each box. Cards will be picked consecutively by a research nurse not otherwise involved in the study. The EXP group will receive aprepitant (EMEND®) in combination with standard anti-emetic treatment and the CTR group will receive standard anti-emetic treatment. All treatment will be given in the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Able to communicate in Swedish
* Diagnosis of lymphoproliferative disease
* Scheduled for myeloablative therapy and autologous stem cell transplantation
* Written informed consent
* Able to swallow oral medications

Exclusion Criteria:

* Nausea at baseline (immediately before start of chemotherapy)
* Gastrointestinal obstruction or active peptic ulcer
* Current illness requiring chronic systemic steroids or requirement for chronic use of antiemetic agent(s)
* Hypersensitivity to any component of the study regimen
* Pregnancy or nursing
* Unrelenting hiccups
* Radiation therapy to pelvis or abdomen within 1 week before or after study day 1
* Psychiatric illness or multi-system organ failure
* Hepatic insufficiency with ASAT, ALAT three times over reference value
* Renal insufficiency with creatinin value three times over reference value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Vomiting and nausea | 7 days
  The proportion of patients with a complete response (no vomiting and/or only mild nausea and no use of rescue therapy) a/ during chemotherapy and b/ in the delayed phase (up to 7 days after end of chemotherapy).

SECONDARY OUTCOMES:
Safety and tolerability of the aprepitant regimen for CINV | 3 weeks
  Possible side effects will be recorded, and all AE:s reported during 3 weeks after the chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Birgegard, MD, PhD, Principal Investigator — University Hospital, Uppsala, Sweden
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden